CLINICAL TRIAL: NCT05392933
Title: Investigation of the Presence of Piriformis Syndrome Accompanying Lumbar Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Yasar Burak Topcu, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IstanbulUC-YasarBurakTOPCU-001
Record Dates: First submitted 2022-03-21; First posted 2022-05-26 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Piriformis Syndrome; Lumbar Radiculopathy
Keywords: Piriformis Syndrome; Lumbar Radiculopathy; Ultrasonography; Diagnostic Injection
MeSH Terms: conditions — Piriformis Muscle Syndrome; Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Piriformis syndrome with lumbar radiculopathy (PSWLR) (Experimental): All patients (n=39) will be evaluated with detailed physical examination and special clinical tests for both lumbar radiculopathy and piriformis syndrome. If patients have lumbar magnetic resonance imaging or electromyography results, they will be recorded to confirm the diagnosis of lumbar radiculopathy. The patients who have the final diagnosis of lumbar radiculopathy and prediagnosis of piriformis syndrome will be evaluated for the pain scores (pain at resting, sitting, standing, lying, at night and during activity) using numeric rating scale. Then, an ultrasound guided piriformis muscle injection will be performed. The patients will be kept under observation for 30 minutes afterwards and the percentage of their pain relief will be recorded. The patients whose pain resolves at least 50% from the baseline after the injection will be diagnosed as piriformis syndrome and will be reevaluated one week and one month after the injection and the changes in the pain scores will be recorded.
  Interventions: Diagnostic Test: Ultrasound guided piriformis muscle lidocaine injection

INTERVENTIONS:
Diagnostic Test: Ultrasound guided piriformis muscle lidocaine injection — Ultrasound guided piriformis muscle (piriformis syndrome) 5 ml %2 lidocaine injection
  Other Names: Ultrasound guided piriformis muscle (piriformis syndrome) diagnostic lidocaine injection

SUMMARY:
Piriformis syndrome is a neuromuscular disorder that is characterized by piriformis muscle tenderness, hip, and leg pain, and may be accompanied by compression or irritation of the sciatic nerve under the piriformis muscle. There are many studies in the literature to establish diagnostic criteria for piriformis syndrome, and there is still no clear consensus on these criteria. However, cases with lumbar radiculopathy were accepted as exclusion criteria in all these studies. The aim of our study is to investigate whether lumbar radiculopathy and piriformis syndrome can coexist. For this reason, a diagnostic piriformis muscle injection under ultrasonography guidance is planned for patients with lumbar radiculopathy who also have a prediagnosis of piriformis syndrome clinically.

DETAILED DESCRIPTION:
Lumbar radiculopathy is a condition in which lumbar spinal nerve roots are affected due to various pathologies. The diagnosis is made clinically by the symptoms and physical examination findings. Most of the time, the diagnosis is supported by imaging methods and electrodiagnostic tests.

Piriformis syndrome is a neuromuscular disorder that is characterized by piriformis muscle tenderness, hip, and leg pain, and may be accompanied by compression or irritation of the sciatic nerve under the piriformis muscle. Similarly, the diagnosis of piriformis syndrome is made clinically based on the patients' history and physical examination. In addition, piriformis muscle injections are an accepted method for the diagnosis of piriformis syndrome. However, the diagnosis of piriformis syndrome is still a controversial issue due to the absence of universally accepted diagnostic criteria, pathognomonic findings, or a gold standard diagnostic method. In this context, many authors have reported that piriformis syndrome is mostly a diagnosis of exclusion. For this reason, the diagnosis of piriformis syndrome is missed in patients with lumbar radiculopathy and these patients may apply to multiple physicians due to their ongoing pain. This can lead to loss of time, financial losses, sensitization and chronic pain in patients and even unnecessary lumbar surgery. Our aim is to investigate whether these two clinical conditions coexist by performing a diagnostic piriformis muscle injection test under ultrasonographic guidance to patients with a diagnosis of lumbar radiculopathy and also with symptoms and signs of piriformis syndrome.

The diagnostic injection test into the piriformis muscle has also been reported to have therapeutic effects. Therefore, the second goal of our study is to investigate the therapeutic effect of piriformis muscle injection in patients diagnosed with lumbar radiculopathy and also piriformis syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18 years
* Having clinical symptoms and signs of L4/L5/S1 radiculopathy which may be supported by imaging and/or electrodiagnostic evaluation
* Having tenderness at the piriformis muscle

Exclusion Criteria:

* Injection history at the lumbar, hip, gluteal region in the last 6 months
* Operation history at the lumbar and/ or hip region
* History of inflammatory rheumatic disease
* History of infectious disease
* History of bleeding disorder
* History of anticoagulation use
* Uncontrolled diabetes mellitus or hypertension
* History of neurological disease
* Being in gestational or lactational period
* Noncompensated chronic heart/liver/renal deficiency, or vascular/tumoral disease
* Active psychiatric disease
* History of allergic reaction to the substance to be applied as local anesthetic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline pain at 30 minutes after piriformis muscle injection | Baseline, 30 minutes after piriformis muscle injection
  After the piriformis muscle injection, the percentage of relief in patient's symptoms will be questioned. It has been reported that 50% or more reduction in the patient's complaints after injecting the local anesthetic agent into the piriformis muscle, with or without steroids, is diagnostic for piriformis syndrome. Therefore, patients with at least 50% reduction in post-injection complaints will be diagnosed with piriformis syndrome.

SECONDARY OUTCOMES:
Change in patient's pain level via Numeric Rating Scale at 1 week and 1 month after injection | Baseline, one week after piriformis muscle injection, one month after piriformis muscle injection
  Before the injection, the participants' pain at resting, sitting, standing, lying, at night, during activity will be assessed by one of the most commonly used pain scale 'numerical rating scale'. It is numeric version of 'visual analog scale' in which the patient selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing "no pain" to '10' representing "pain as bad as you can imagine". One week after the injection, the participant's pain while resting, walking, sitting, lying down and at night will be evaluated with a numerical rating scale and the change in pain scores will be evaluated. Similarly, the change in pain scores during the same activities one month after the injection will also be evaluated. In this way, the amount of relief that may be provided via the piriformis muscle injection in patients having lumbar radiculopathy and piriformis syndrome in short and medium terms will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Yasar Burak Topcu, Principal Investigator — Istanbul University - Cerrahpasa; Tugce Ozekli Misirlioglu, Study Director — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tarulli AW, Raynor EM. Lumbosacral radiculopathy. Neurol Clin. 2007 May;25(2):387-405. doi: 10.1016/j.ncl.2007.01.008. PMID 17445735
- [Background] Bogduk N. On the definitions and physiology of back pain, referred pain, and radicular pain. Pain. 2009 Dec 15;147(1-3):17-9. doi: 10.1016/j.pain.2009.08.020. Epub 2009 Sep 16. No abstract available. PMID 19762151
- [Background] Probst D, Stout A, Hunt D. Piriformis Syndrome: A Narrative Review of the Anatomy, Diagnosis, and Treatment. PM R. 2019 Aug;11 Suppl 1:S54-S63. doi: 10.1002/pmrj.12189. Epub 2019 Jul 22. PMID 31102324
- [Background] Michel F, Decavel P, Toussirot E, Tatu L, Aleton E, Monnier G, Garbuio P, Parratte B. Piriformis muscle syndrome: diagnostic criteria and treatment of a monocentric series of 250 patients. Ann Phys Rehabil Med. 2013 Jul;56(5):371-83. doi: 10.1016/j.rehab.2013.04.003. Epub 2013 Apr 25. PMID 23684470
- [Background] Siddiq MA, Hossain MS, Uddin MM, Jahan I, Khasru MR, Haider NM, Rasker JJ. Piriformis syndrome: a case series of 31 Bangladeshi people with literature review. Eur J Orthop Surg Traumatol. 2017 Feb;27(2):193-203. doi: 10.1007/s00590-016-1853-0. Epub 2016 Sep 19. PMID 27644428
- [Background] Hopayian K, Song F, Riera R, Sambandan S. The clinical features of the piriformis syndrome: a systematic review. Eur Spine J. 2010 Dec;19(12):2095-109. doi: 10.1007/s00586-010-1504-9. Epub 2010 Jul 3. PMID 20596735
- [Background] Fishman LM, Dombi GW, Michaelsen C, Ringel S, Rozbruch J, Rosner B, Weber C. Piriformis syndrome: diagnosis, treatment, and outcome--a 10-year study. Arch Phys Med Rehabil. 2002 Mar;83(3):295-301. doi: 10.1053/apmr.2002.30622. PMID 11887107
- [Background] Jankovic D, Peng P, van Zundert A. Brief review: piriformis syndrome: etiology, diagnosis, and management. Can J Anaesth. 2013 Oct;60(10):1003-12. doi: 10.1007/s12630-013-0009-5. Epub 2013 Jul 27. PMID 23893704
- [Background] Miller TA, White KP, Ross DC. The diagnosis and management of Piriformis Syndrome: myths and facts. Can J Neurol Sci. 2012 Sep;39(5):577-83. doi: 10.1017/s0317167100015298. PMID 22931697
- [Background] Papadopoulos EC, Khan SN. Piriformis syndrome and low back pain: a new classification and review of the literature. Orthop Clin North Am. 2004 Jan;35(1):65-71. doi: 10.1016/S0030-5898(03)00105-6. PMID 15062719
- [Background] Misirlioglu TO, Akgun K, Palamar D, Erden MG, Erbilir T. Piriformis syndrome: comparison of the effectiveness of local anesthetic and corticosteroid injections: a double-blinded, randomized controlled study. Pain Physician. 2015 Mar-Apr;18(2):163-71. PMID 25794202
- [Background] Terlemez R, Ercalik T. Effect of piriformis injection on neuropathic pain. Agri. 2019 Nov;31(4):178-182. doi: 10.14744/agri.2019.34735. PMID 31741344
- [Background] Lauder TD. Physical examination signs, clinical symptoms, and their relationship to electrodiagnostic findings and the presence of radiculopathy. Phys Med Rehabil Clin N Am. 2002 Aug;13(3):451-67. doi: 10.1016/s1047-9651(02)00006-2. PMID 12380545